CLINICAL TRIAL: NCT04227405
Title: TOGETHER: A Couple's Model to Enhance Relationships and Economic Stability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding agency (Administration of Children and Families, US Department of Health and Human Services) discontinued the local evaluation
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Maryland, Baltimore (Other); Family Services, Inc. (Industry); The SkillSource Group, Inc. (Other); AVAR Consulting, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-960
Record Dates: First submitted 2018-05-09; First posted 2020-01-13 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-07

CONDITIONS: No Condition

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group of couples will receive no intervention
- Intervention (Experimental): Intervention group of couples received the intervention: case management (connection to community services), 20 hour pscycho-educational workshop on communication, conflict resolution, problem-solving, stress management, and financial management, booster session, and employment support services if needed
  Interventions: Behavioral: Connection to community services through case management; Behavioral: TOGETHER Workshop; Behavioral: Employment Support Services

INTERVENTIONS:
Behavioral: Connection to community services through case management — Case managers met with couple and conduct a needs assessment for the couple and their family. Then they developed an Individual and Couple Development Plan to take care of those needs, usually by accessing community services. Case managers met every 5 weeks with the couple to check on progress toward meeting the goals of the plan and assess for the present of any new needs.
  Arms: Intervention
Behavioral: TOGETHER Workshop — Couples were required to participate in a 20 hour workshop (8 sessions of 2 1/2 hours each)in groups of 3 to 8 couples. These groups were facilitated by a financial expert and a couples' expert. The workshop is interdisciplinary and psycho-educational. Couples learn about skills to improve their communication about stress and money problems, conflict resolution, individual and couple stress management in general and about money stress in particular, and financial management
  Arms: Intervention
Behavioral: Employment Support Services — Only for those participants that were in need of employment support services. If the needs assessment conducted by the case manager indicated an employment or career need. After completion of the TOGETHER workshop, an employment case manager met with the participant, conducted an employment needs assessment and connected the participant with a workforce agency or one-stop employment centers. After doing so, the employment case manager followed through the various steps that the participant had to complete as part of the employment services for a period of 6 months
  Arms: Intervention

SUMMARY:
The current study sought to evaluate an intervention to promote healthy couple relationships and economic stability and mobility for low-income couples living in Northern Virginia (VA) and Montgomery and Prince George's Counties (MD). The approach proposed integrated two components:(1) a 20-hour evidence-informed couple group workshop called TOGETHER that integrates relationship and financial education, followed by an optional three-hour booster session three months after TOGETHER workshop and (2) case management (assessment of participant needs, development of Individual and Couple Development Plan(ICDP), referrals for social and mental health services, and referrals and coordination with job and career enhancement services, linking and coordination of all services as needed). The 20-hour workshop was offered in 8 sessions facilitated by couple and financial experts. The effectiveness of the program was evaluated through a randomized control trial in which couples were randomly assigned to a control group (n=147) or an intervention group (n=145). The control group received no intervention but a three-hour financial workshop after the last assessment was completed whereas the intervention couples participated in the 20-hour interventions and received case management. An independent local evaluator(AVAR, Consulting) participated in the design, implementation, and most of the data analysis. Participants had to be at least 18 years-old, living together for at least a year, and had no severe domestic violence issues, or untreated substance abuse or severe psychiatric disorders. If both partners were retired, couples were excluded from participation. Couples participated in an intake and enrollment meeting and were randomly assigned by a computer generated system to either the intervention or control group. Couples in both groups completed three sets of self-report measures: (1)Pre-test in first workshop session or at intake for control couples, (2)post-test in the last workshop session, or 8 weeks after the pre-test for control couples, and (3)follow-up six months after the post-test. After the six-month follow-up assessment, participation in the program was concluded. The study was largely funded by a Healthy Marriage and Responsible Fatherhood grant awarded by the Administration of Children and Families.

DETAILED DESCRIPTION:
The current project sought to promote healthy couple relationships and economic stability and mobility for low-income couples living in Northern Virginia (VA) and Montgomery and Prince George's Counties (MD) This project was funded by the Administration for Children and Families (ACF) under the Healthy Marriage and Responsible Fatherhood (HMRF) program from the beginning of the study until May 10, 2018. As of May 10, 2018 ACF continued to fund the intervention component but data collection and analysis for couples that had been randomized by then and continued to receive services and to complete assessments were funded by Virginia Polytechnic Institute and State University. The evaluation plan that included a randomized control trial (RCT) and was approved of by ACF for years 2016, 2017, and 2018 until the local evaluation was discontinued by ACF included the enrollment of 720 couples, out of which 360 couples would be randomly assigned to the intervention group and 360 couples to a control group. However, due to the unexpected termination of funding for the local evaluation, the program was evaluated with 292 couples (145 intervention group couples and 147 control group couples).

This project was developed and conducted by Project Director, Mariana Falconier, Ph.D. at Virginia Tech and Associate Director until December, 2018 and since then at the University of Maryland (UMD), and Jinhee Kim, Ph.D. at UMD. UMD was a subawardee of Virginia Tech. Virginia Tech subcontracted with SkillSource Group, Inc. for delivery of employment services and University of Maryland contracted with Family Services, Inc. for delivery of workshop services. ACF required the grantee to have an independent local evaluator and for that purpose Virginia Tech contracted with AVAR Consulting, involved in the implementation and outcome evaluations until August 31, 2018. Additional analyses were conducted by D. Mark Lachowicz from UMD.

Our approach integrated two components (1) a 20-hour evidence-informed couple group program called TOGETHER workshop that integrates relationship education and financial literacy skills and (2) case management (assessment of participant needs, development of Individual and Couple Development Plan, referrals for community services, and referrals and coordination with job and career enhancement services).

Short-term outcomes of this project's core intervention were expected immediately after completion of the last session of the TOGETHERR workshop whereas medium-term outcomes were anticipated six months after that last session. Expected measurable outcomes among program participants for objective 1 (improved personal well-being) included increased frequency of positive stress management, reduced psychological distress, decreased financial stress. Expected measurable outcomes for objective 2 (improved couple's relationship skills) included increased frequency of positive communication behaviors, increased frequency of positive conflict management behaviors, increased frequency of positive dyadic stress management, increased frequency of conjoint problem solving behaviors, increased satisfaction with couple's relationship, and increased comfort with financial styles and roles. Expected measurable outcomes for objective 3 (improved parenting and co-parenting) included increased frequency of positive parenting behaviors, increased closeness to children, and increased satisfaction with co-parenting. Expected measurable outcomes for objective 4 (improved financial literacy and capability) include increased financial literacy skills, increased financial self-efficacy, decreased use of alternative financial services, and increased financial management behaviors. Finally, expected measurable outcomes for objective 5 (improved employability, job placement, and retention) include decreased perceived barriers to employability, increased intentions and motivations for work, increased confidence in job skills, and increased employability, employment status, and retention. These outcomes were expected by comparing the intervention and control group outcomes in the RCT.

Outcomes were evaluated through self-report measures provided ACF and additional standardized measures selected by the Project Director and Associated Project Director. Measures were completed at baseline, 8 weeks after, and six-month follow up. Couples received gift cards for survey completion.

TARGET POPULATION Low income couples in Northern Virginia (VA) and Prince George's County and Montgomery County, Maryland (MD) but all couples were if they met the eligibility criteria: Living together at least a year, 18 years or older, and English-speaking. Exclusion criteria included both partners being retired, physical domestic violence or feeling unsafe with partner in the last six months, untreated severe psychiatric disorder or/and severe untreated substance abuse disorder. Couples could participate as long as both partners consent to be part of the program.

RECRUITMENT Recruitment activities began on June 1, 2016 and included advertising through social media, distributing flyers, brochures, and posters and/or giving presentation in schools, churches and various community agencies. The program was also advertised through its own website.

DATABASES The funding agency ACF requires all HMRF grantees to enter information into a secure system called the Information, Family Outcomes, Reporting, and Management system (nFORM) regarding program operations, services,a nd participants' contract information and demographics. ACF required grantees to collect their outcome measures through nFORM and the researches added standardized self-report instrument to be collected through Qualtrics. Both nFORM and Qualtrics measures were used for the RCT. A database called Participant Tracking System (PTS) was developed for automated randomization and entering needs assessments and ICDPs.

PROCEDURES Individuals interested in participating in the program could contact us in person or by phone. Program staff collected contact information, described the program and the potential compensation, asked screening questions to each partner if both partners were available. Otherwise, the program staff collected information from the only partner that was present. Eligible participants that provided consent were scheduled for an Intake and Enrollment (IE) meeting with the case managers.

The first part of the IE meeting lasted 60 minutes. During the meeting, the case manager (a) described the program and obtained voluntary, informed written consent for program participation from both partners; (b) conducted a 10-minute formal assessment of domestic violence with each partner individually (couples at risk were referred to outside agency); (c) enrolled participants in nFORM; (d) assigned couples to intervention or control group through an automated system of randomization; (f) provided orientation about program procedures; and (g) directed couples to complete the nFORM applicant characteristics survey and a Qualtrics demographic information survey in a tablet The second part of the IE meeting was different for intervention and control couples. For intervention couples (90 minutes), the case manager described the services, conducted a Needs Assessment (areas: Health care, employment, housing, childcare, education, legal needs, finances, transportation, food, relationships, mental health, alcohol abuse, and substance abuse), scheduled the individual and couple development plan (ICDP) meeting and case management progress and exit meetings, and enrolled couples in one of the eight-week TOGETHER workshops and a three-hour booster session (three months the TOGETHER workshop. During part II (90 minutes) for control couples completed pre-test surveys including the Pre-Program Survey (nFORM) and Pre-test Assessment (Qualtrics).

Eight weeks after the IE meeting, control couples would meet with the case manager in a program location and complete the Post Program Survey in nFORM and the Post-test Assessment in Qualtrics (90 minutes) and received gift cards. Questionnaires mailed for those unable to attend. Six months later couples were invited to complete the follow-up survey in Qualtrics (90 minutes) before the beginning of the Financial Literacy Workshop (FLW). They received gift cards. If unable to attend, paper surveys were mailed. FLW was a three-hour financial management class to improve financial management knowledge and skills based on Money Smart curriculum.

INTERVENTION COUPLES

1. TOGETHER WORKSHOP TOGETHER workshop is a 20-hour psycho-educational program that integrates relationship and financial education. TOGETHER was developed by Dr. Mariana Falconier (PI) and the late Dr. Hayhoe as part of the emerging interdisciplinary field that integrates relationship education with financial education (Falconier, 2015). TOGETHER adapted the Couples' Coping Enhancement Training (CCET; Bodenmann & Shantinah, 2004), whose effectiveness in improving stress management, communication, and relationship satisfaction has been supported in various studies (e.g., Bodenmann & Shantinath, 2004), to financial stress. TOGETHER aims at reducing financial stress and improving relationship functioning by providing couples with knowledge and skills on individual and couple's stress management, communication, conflict resolution, problem-solving, and financial management. The TOGETHER workshop has 9 modules and is designed to be delivered in groups of four to eight couples: 8 weekly sessions of 2.5 hours each. Each session is co-led by two facilitators: a financial counselor and a couple therapist. Each session includes a warm-up activity, brief review of past session content and homework, presentation and practice of new content, summary of all contents covered in the session, and assignment of new homework. The TOGETHER curriculum has been pilot tested and results have been published in 2015 in the Journal of Marital and Family Therapy.

   Program Modules Introduction to program Module 1: Understanding Stress and Money Stress Module 2: Managing* Stress and Money Stress by Yourself Module 3: Communicating Stress and Money Stress to Your Partner Module 4: Managing Stress and Money Stress with Your Partner Module 5: Communicating Effectively and Learning to Talk about Money Module 6: Clarifying Financial Roles and Expectations Module 7: Improving Money Management Skills Module 8: Credit and Risk Management Module 9: Improving Financial Problem-Solving Skills Thirty workshops were offered between July 1, 2016 and May 10, 2018. Out of the 145 couples assigned to the intervention group, 106 couples started the workshop. The rest of the couples could not attend any of the available workshops due to schedule conflicts. At the end of each session participants completed a 2 minute-session evaluation (last session survey also includes questions about the overall workshop) and a 2-minute homework evaluation.. At the first TOGETHER session, couples completed the Pre Program Survey (nFORM) and the Pre-test Assessment (Qualtrics) (total = 90 minutes) on a tablet before the session began. Couples absent in the first session were mailed paper surveys. After the last (eighth) TOGETHER session, couples completed on site the Post Program Survey (nFORM) and the Post-test Assessment (Qualtrics) (90 minutes) on tables or were mailed paper surveys if they failed to attend.
2. CASE MANAGEMENT One week after the first workshop session, intervention couples partook in an Individual and Couple Development Plan (ICDP) meeting with the assigned case. Based on the information collected in the Needs Assessment during the IE meeting, the case manager created an ICDP with the couple that included goals, action steps, potential barriers, and referrals to community services (i.e., housing, TANF, health care, mental health services, etc.). If the ICDP included a goal related employment/career a first meeting was scheduled for that partner with an employment case manager to receive services at either the SkillSource Group, Inc. or a federally funded employment agency in Maryland. The present study provided funding for (a) employment services for those participants that did not meet eligibility criteria to receive services funded through the Workforce Innovation and Opportunity Act (WIOA) or other state and local funding in those agencies.

   After the ICDP meeting, intervention couples met with the case manager for their five progress monthly meetings in order to check participants' progress towards goals, barriers, safety, program issues, and modifications to ICDP. There was an exit meeting with the case manager 6 months after the last TOGETHER workshop session during which couples completed the six-month follow-up survey. If unable to attend, paper surveys were mailed.
3. INCENTIVES FOR WORKSHOP ATTENDANCE At the third progress meeting, case managers provided the attendance incentives for the TOGETHER workshop.
4. BOOSTER SESSION Intervention couples were invited to an optional 3- hour booster session (abbreviated version of workshop content) three months after completing the last session of TOGETHER workshop.
5. FIDELITY Facilitators received a 25-hour training in the program, a biweekly one-hour group supervision with the curriculum developers, were observed by the curriculum developers and the local evaluators staff. Facilitators also completed jointly a checklist to report on the extent to which they completed the scheduled activities, met all session objectives, used all materials as outlined in the manual, and spent the time as planned.

A checklist was developed to assess the extent to which case managers were implementing the case management protocol.

ELIGIBILITY:
Inclusion Criteria

* Lliving together for at least a year
* Being at least 18 years
* English speaking.

Exclusion criteria:

* Current physical domestic violence and/ or feeling unsafe to participate with your partner in a psycho-educational group in the last twelve months
* Current diagnosis of a severe psychiatric disorder that required hospitalization in the last 12 months
* Cognitive impairment that prevent comprehension of materials and participation in a psycho-educational group
* Severe untreated substance abuse disorder
* Both partners fully retired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana K Falconier, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (3):
- United States (3):
  - University of Maryland, College Park, Maryland
  - Family Services, Inc., Gaithersburg, Maryland
  - Virginia Tech Northern Virginia Center, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falconier MK. Together - a couples' program to improve communication, coping, and financial management skills: development and initial pilot-testing. J Marital Fam Ther. 2015 Apr;41(2):236-50. doi: 10.1111/jmft.12052. Epub 2014 Jun 9. PMID 24910157
- See also: Program's Website — http://www.togetherprogram.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Intervention group of couples received the intervention: case management (connection to community services), 20 hour pscycho-educational workshop on communication, conflict resolution, problem-solving, stress management, and financial management, booster session, and employment support services if needed
  Connection to community services through case management: Case managers met with couple and conduct a needs assessment for the couple and their family. Then they developed an Individual and Couple Development Plan to take care of those needs, usually by accessing community services. Case managers met every 5 weeks with the couple to check on progress toward meeting the goals of the plan and assess for the present of any new needs.
  TOGETHER Workshop: Couples were required to participate in a 20 hour workshop (8 sessions of 2 1/2 hours each)in groups of 3 to 8 couples. These groups were facilitated by a financial expert and a couples' expert. The workshop is interdisciplinary
Period: Enrollment - Time 1 PreTest
Arm/Group | Control Group | Intervention
Started | 294 | 290
Completed | 268 | 212
Not Completed | 26 | 78
Not completed — Schedule conflict /uninterested/Barriers | 26 | 78
Period: Time 1 PreTest - Time 2 PostTest
Arm/Group | Control Group | Intervention
Started | 268 | 212
Completed | 186 | 144
Not Completed | 82 | 68
Not completed — Conflict schedule/uninterested/barriers | 82 | 68
Period: Time 2 PostTest - Time 3 Followup
Arm/Group | Control Group | Intervention
Started | 186 | 144
Completed | 118 | 96
Not Completed | 68 | 48
Not completed — Uninterested-Barriers to participation | 68 | 48

BASELINE CHARACTERISTICS:
Population: This study was terminated and the PI no longer works for the sponsor institution, nor is the data accessible to Virginia Tech as it was removed from the institution in the care of the PI. What has been provided in the baseline analysis is all of the data available.
Groups:
- Intervention: Intervention group of couples received the intervention: case management (connection to community services), 20 hour pscycho-educational workshop on communication, conflict resolution, problem-solving, stress management, and financial management, booster session, and employment support services if needed
  Connection to community services through case management: Case managers met with couple and conduct a needs assessment for the couple and their family. Then they developed an Individual and Couple Development Plan to take care of those needs, usually by accessing community services. Case managers met every 5 weeks with the couple to check on progress toward meeting the goals of the plan and assess for the present of any new needs.
  TOGETHER Workshop: Couples were required to participate in a 20 hour workshop (8 sessions of 2 1/2 hours each)in groups of 3 to 8 couples. These groups were facilitated by a financial expert and a couples' expert. The workshop is interdisciplinary and p
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention | Total
Number analyzed (Participants) | 294 | 290 | 584
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 292 | 287 | 579
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.90 (10.79) | 37.93 (10.53) | 38.93 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 148 | 298
  Male | 144 | 142 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 38 | 68
  Not Hispanic or Latino | 247 | 235 | 482
  Unknown or Not Reported | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 4 | 11
  Asian | 11 | 29 | 40
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 170 | 144 | 314
  White | 85 | 94 | 179
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 17 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 294 | 290 | 584

OUTCOME MEASURES:

1. Primary Outcome: Information, Family Outcomes, Reporting, and Management (nFORM)- Baseline/Pretest (Time1)
Description: nFORM survey was developed by Mathematica. Subscales: Depression (4 items; Range: 4-20); Anxiety (2 items; Range: 2-10); Positive conflict management (7 items; Range: 7-28); Negative conflict management (5 items; Rrange: 5-20); Emotional abuse (2 items; Range: 2-8); Conflict management Satisfaction (1 item; Range: 1-3); Relationship quality (5 items; Range:5-20); Time with partner (3 items; Range: 3-12); Relationship Satisfaction (1 item; Range: 1-3); Parenting stress (1 item; Scale range: 1-4); Banking (3 items; Range: 0-3); Difficulty to pay bills (1 item; Scale range: 1 - 4); Relationship Commitment (1 item; Range: 1); Budgeting (1 item; Range: 0-1). Range is Scale Range. Higher scores means higher levels on that variable.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Pre-test/Baseline (Time 1) (Completed in first workshop session for Intervention Group and int the Intake and Enrollment Meeting for the Control Group)
Population: 294 individuals (147 couples) were assigned to control group but only 268 indiividuals (134 couples) completed the pre-test survey.
  290 individuals (145 couples) were assigned to the intervention group but only 212 individuals (106 couples) completed the pre-test survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Depression | 7.44 (2.95) | 8.33 (3.24)
  Anxiety | 4.31 (1.77) | 5.18 (1.85)
  Positive Conflict Management | 21.27 (3.93) | 20.61 (4.17)
  Negative Conflict Management | 12.6 (3.75) | 13.39 (3.83)
  Emotional Abuse | 4.36 (1.84) | 4.61 (1.89)
  Conflict Management Satisfaction Scale | 2 (0.71) | 1.83 (0.71)
  Relationship Quality | 16.12 (3.41) | 15.84 (3.03)
  Time with Partner | 9.97 (2.20) | 9.87 (2.11)
  Relationship Satisfaction | 2.32 (0.72) | 2.25 (0.69)
  Parenting Stress | 2.63 (0.98) | 2.64 (0.85)
  Banking | 1.65 (0.65) | 1.74 (0.56)
  Difficulty to pay bills | 2.29 (0.96) | 2.4 (1)
  Relationship Commitment | 3.46 (0.74) | 3.58 (0.64)
  Budgeting | 0.41 (0.49) | 0.45 (0.5)

2. Primary Outcome: Information, Family Outcomes, Reporting, and Management (nFORM)- Post-test at 8 Weeks After Pre-test (Time2)
Description: nFORM survey was developed by Mathematica. Subscales: Depression (4 items; Range: 4-20); Anxiety (2 items; Range: 2-10); Positive conflict management (7 items; Range: 7-28); Negative conflict management (5 items; Rrange: 5-20); Emotional abuse (2 items; Range: 2-8); Conflict management Satisfaction (1 item; Range: 1-3); Relationship quality (5 items; Range:5-20); Time with partner (3 items; Range: 3-12); Relationship Satisfaction (1 item; Range: 1-3); Parenting stress (1 item; Scale range: 1-4); Banking (3 items; Range: 0-3); Difficulty to pay bills (1 item; Scale range: 1 - 4); Relationship Commitment (1 item; Range: 1-4); Budgeting (1 item; Range: 0-1). Range is Scale Range. Higher scores means higher levels on that variable.
Time Frame: Post-test (8 weeks after pre-test/Time1)
Population: 294 individuals (147 couples) were assigned to control group but only 186 indiividuals (93 couples) completed the pre-test survey.
  290 individuals (145 couples) were assigned to the intervention group but only 144 individuals (72 couples) completed the pre-test survey
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Depression | 6.92 (3) | 7.48 (3.1)
  Anxiety | 4.28 (1.7) | 4.64 (1.71)
  Positive Conflict Management | 21.91 (3.51) | 22.09 (3.9)
  Negative Conflict Management | 11.69 (3.98) | 11.96 (3.89)
  Emotional Abuse | 3.85 (1.75) | 3.90 (1.77)
  Conflict Management Satisfaction | 2.2 (0.69) | 2.16 (0.66)
  Relationship Quality | 16.39 (3.35) | 16.71 (2.86)
  Time with Partner | 10.16 (2.08) | 9.97 (1.93)
  Relationship Satisfaction | 2.43 (0.66) | 2.5 (0.62)
  Parenting Stress | 2.49 (0.89) | 2.60 (0.82)
  Banking | 1.73 (0.6) | 1.74 (0.56)
  Difficulty to Pay Bills | 2.1 (0.81) | 2.31 (1)
  Relationship Commitment | 3.44 (0.72) | 3.65 (0.61)
  Budgeting | 0.64 (0.51) | 0.71 (0.46)
Statistical Analysis 1: Comparison: Control Group; Change between pre-test and post-test for the Positive Conflict Management subscale using multilevel modeling; Test type: Superiority; p > .05, Multilevel modeling — The Benjamini-Hochberg method (1995) was used for adjusting p values for multiple comparisons as recommended by What Works Clearinghouse for controlling the false discovery rate for studies that have multiple outcome variables; Slope = 0.24, Standard Error of Mean 0.23 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change between pre-test and post-test for the Positive Conflict Management subscale using multilevel modeling; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.59, Standard Error of Mean 0.29 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Positive Conflict Management subscale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.35, Standard Error of Mean 0.36 — The increase from pre-test to post-test in the intervention group is significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 4: Comparison: Control Group; Change from pre-test to post-test in Negative Conflict Management for the Control Group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.47, Standard Error of Mean 0.23 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from pre-test to post-test in the Negative Conflict Management subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -1.48, Standard Error of Mean 0.29 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Negative Conflict Management subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -1.00, Standard Error of Mean 0.36 — The expected decrease from pre-test to post-test in the intervention group is significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 7: Comparison: Control Group; Changes in the Relationship Quality subscale from Pre-test to post-test in the control group; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.33, Standard Error of Mean 0.14 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Changes in the Relationship Quality Subscale from pretest to posttest in the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.86, Standard Error of Mean 0.17; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Relationship Qualitty subscale; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.53, Standard Error of Mean 0.22; The expected increase from pre-test to post-test in the intervention group is significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 10: Comparison: Control Group; Changes from pre-test to posttest in the Emotional Abuse subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.32, Standard Error of Mean 0.11 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Changes from pre-test to posttest in the Emotional Abuse subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.71, Standard Error of Mean 0.13; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Emotional Abuse subscale; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.39, Standard Error of Mean 0.16; The expected decrease from pre-test to post-test in the intervention group is significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 13: Comparison: Control Group; Changes from pre-test to posttest in the Relationship Satisfaction subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.02, Standard Error of Mean 0.04; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 14: Comparison: Intervention; Changes from pre-test to posttest in the Relationship satisfaction subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.28, Standard Error of Mean 0.05 — The expected increase from pre-test to post-test in the intervention group is significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 15: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Relationship Satisfactionn subscale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.26, Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 16: Comparison: Control Group; Changes from pre-test to posttest in the Relationship Commitment subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.05, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 17: Comparison: Intervention; Changes from pre-test to posttest in the Relationship Commitment subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.22, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 18: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Relationship Commitment subscale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.27, Standard Error of Mean 0.07 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 19: Comparison: Control Group; Changes from pre-test to posttest in the Depression subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment in p value; Slope = -0.7, Standard Error of Mean 0.17 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 20: Comparison: Intervention; Changes from pre-test to posttest in the Depression subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment in p value; Slope = -0.81, Standard Error of Mean 0.21; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 21: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Depression subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.11, Standard Error of Mean 0.26 — Changes from pre-test to post-test in the intervention group were not significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 22: Comparison: Control Group; Changes from pre-test to posttest in the Anxiety subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.26, Standard Error of Mean 0.10 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 23: Comparison: Intervention; Changes from pre-test to posttest in the Anxiety subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment in p value; Slope = -0.41, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 24: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Anxiety subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.15, Standard Error of Mean 0.16 — Changes from pre-test and post-test in the intervention group were not significantly different from the change from pre-test and post-test in the control group
Statistical Analysis 25: Comparison: Control Group; Changes from pre-test to posttest in Budgeting subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.11, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 26: Comparison: Intervention; Changes from pre-test to posttest in the Budgeting subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.23, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 27: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Budgeting subscale; Test type: Superiority; p < .10, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.12, Standard Error of Mean 0.05 — Changes from pre-test to follow-up in the intervention group were not significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 28: Comparison: Control Group; Changes from pre-test to posttest in the Difficulties to Pay Bills subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling — No adjustment in p value; Slope = -0.1, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 29: Comparison: Intervention; Changes from pre-test to posttest in the Difficulties to Pay Bills subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment in p value; Slope = -0.21, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 30: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Difficulties to Pay Bills subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.12, Standard Error of Mean 0.08; Changes from pre-test to post-test in the intervention group were not significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 31: Comparison: Control Group; Changes from pre-test to posttest in Time with Partner subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = 0.11, Standard Error of Mean 0.11 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 32: Comparison: Intervention; Changes from pre-test to posttest in Time with Partner subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment in p value; Slope = 0.28, Standard Error of Mean 0.13 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 33: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Time with Partner subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = 0.16, Standard Error of Mean 0.17 — Changes from pre-test to pos-test in the intervention group were not significantly different from the change from pre-test to pos-test in the control group
Statistical Analysis 34: Comparison: Control Group; Change from pre-test to post-test in banking subscale for control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = 0.03, Standard Error of Mean 0.04 — Positive values indicate an increase whereas a negative value indicates a decrease
Statistical Analysis 35: Comparison: Intervention; Change from pre-test to post-test in banking subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = 0.04, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 36: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Banking subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = 0.02, Standard Error of Mean 0.06; Changes from pre-test to post-test in the intervention group were not significantly different from the change from pre-test to pos-test in the control group
Statistical Analysis 37: Comparison: Control Group; Change from pre-test to post-test in parenting stress subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.05, Standard Error of Mean 0.07 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 38: Comparison: Intervention; Change from pre-test to post-test in parenting stress subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.09, Standard Error of Mean 0.08 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 39: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Parenting stresss subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.05, Standard Error of Mean 0.11 — Changes from pre-test to post-test in the intervention group were not significantly different from the change from pre-test to pos-test in the control group
Statistical Analysis 40: Comparison: Control Group; Change from pre-test to post-test in conflict management satisfaction subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.14, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 41: Comparison: Intervention; Change from pre-test to post-test in conflict management satisfaction subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.32, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 42: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Conflict Management Satisfaction subscale; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.19, Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 3]

3. Primary Outcome: Information, Family Outcomes, Reporting, and Management (nFORM)- Six-month Follow-up (Time3)
Description: nFORM survey was developed by Mathematica.Subscales: Depression (4 items; Range: 4-20); Anxiety (2 items; Range: 2-10); Positive conflict management (7 items; Range: 7-28); Negative conflict management (5 items; Rrange: 5-20); Emotional abuse (2 items; Range: 2-8); Conflict management Satisfaction (1 item; Range: 1-3); Relationship quality (5 items; Range:5-20); Time with partner (3 items; Range: 3-12); Relationship Satisfaction (1 item; Range: 1-3); Parenting stress (1 item; Scale range: 1-4); Banking (3 items; Range: 0-3); Difficulty to pay bills (1 item; Scale range: 1 - 4); Relationship Commitment(1 item; Range: 1-4); Budgeting (1 item; Range: 0-1). Range is Scale Range. Higher scores means higher levels on that variable.
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: 294 individuals (147 couples) were assigned to control group but only 118 indiividuals (59 couples) completed the pre-test survey.
  290 individuals (145 couples) were assigned to the intervention group but only 96 individuals (48 couples) completed the pre-test survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Depression | 6.74 (3.13) | 7.41 (3.03)
  Anxiety | 4.25 (1.81) | 4.64 (1.69)
  Positive Conflict Management | 22 (4.19) | 22.78 (3.63)
  Negative Conflict Management | 11.56 (4.4) | 11.62 (3.9)
  Emotional Abuse | 3.95 (1.96) | 3.87 (1.82)
  Conflict Management Satisfaction | 2.15 (0.73) | 2.17 (0.7)
  Relationship Quality | 16.11 (3.69) | 17.08 (2.74)
  Time with Partner | 9.85 (2.43) | 10.39 (1.65)
  Relationship Satisfaction | 2.41 (0.73) | 2.49 (0.65)
  Parenting Stress | 2.36 (1.00) | 2.50 (.82)
  Banking | 1.79 (0.54) | 1.93 (0.44)
  Difficulty to Pay Bills | 2.17 (0.85) | 2.04 (0.79)
  Relationship Commitment | 3.47 (0.76) | 3.62 (0.66)
  Budgeting | 0.85 (0.36) | 0.93 (0.26)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to Follow-up in the Positive Conflict Management subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.18, Standard Error of Mean 0.28 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to Follow-up in the Positive Conflict Management subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.53, Standard Error of Mean 0.35 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up n the Positive Conflict Management subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.35, Standard Error of Mean 0.44 — Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Positive Conflict Management subscale
Statistical Analysis 4: Comparison: Control Group; Changes from pre-test to Follow-up in the Negative Conflict subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.41, Standard Error of Mean 0.28 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Changes from pre-test to Follow-up in the Negative Conflict Manageement subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -1.4, Standard Error of Mean 0.34; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up n the Negative Conflict Management subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.99, Standard Error of Mean 0.44 — The expected decrease from pre-test to follow-i[in the intervention group is significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 7: Comparison: Control Group; Changes from pre-test to Follow-up in the Relationship Quality subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.41, Standard Error of Mean 0.17 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Changes from pre-test to Follow-up in the Relationship Quality subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.91, Standard Error of Mean 0.21 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up n the Relationship Quality subscale; Test type: Superiority; p < .10, Multilevel modeling — The Benjamini-Hochberg method (1995) was used for adjusting p values for multiple comparisons as recommended by What Works Clearinghouse for controlling the false discovery rate for studies that have multiple outcome variables. Pvalue set at <.05; Slope = 0.5, Standard Error of Mean 0.26 — The expected increase from pre-test to follow-up in the intervention group is not significantly (p > .05) different from the change from pre-test to follow-up in the control group
Statistical Analysis 10: Comparison: Control Group; Changes from pre-test to Follow-up in the Emotional Abuse subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.31, Standard Error of Mean 0.13 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Changes from pre-test to Follow-up in the Emotional Abuse subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.71, Standard Error of Mean 0.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Emotional Abuse subscale; Test type: Superiority; p < .10, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.41, Standard Error of Mean 0.2 — The expected decrease from pre-test to follow-up in the intervention group is not significantly (p > .05) different from the change from pre-test to follow-up in the control group
Statistical Analysis 13: Comparison: Control Group; Changes from pre-test to Follow-up in the Relationship subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.03, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 14: Comparison: Intervention; Changes from pre-test to Follow-up in the Relationship Satisfaction subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.29, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 15: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Relationship Satisfaction subscale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.26, Standard Error of Mean 0.07 — The expected increase from pre-test to follow-up in the intervention group is significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 16: Comparison: Control Group; Changes from pre-test to Follow-up in the Relationship Commitment subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.08, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 17: Comparison: Intervention; Changes from pre-test to Follow-up in the Relationship Commitment subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.24, Standard Error of Mean 0.07 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 18: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Relationship Commitment subscale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.32, Standard Error of Mean 0.09 — [estimate comment as in outcome 3, analysis 15]
Statistical Analysis 19: Comparison: Control Group; Changes from post-test to Follow-up in the Positive Conflict Management subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.06, Standard Error of Mean 0.1 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 20: Comparison: Intervention; Changes from post-test to Follow-up in the Positive Conflict Management subscale for th eintervention group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.06, Standard Error of Mean 0.1 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 21: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Positive Conflict Management subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0, Standard Error of Mean 0.14 — Changes from post-test to follow-up in the intervention group were not significantly different from the change from post-test to follow-up in the control group
Statistical Analysis 22: Comparison: Control Group; Changes from post-test to Follow-up in the Negative Conflict Management subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.06, Standard Error of Mean 0.1 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 23: Comparison: Intervention; Changes from post-test to Follow-up in the Negative Conflict Management subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.08, Standard Error of Mean 0.1 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 24: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Negative Conflict Management subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.01, Standard Error of Mean 0.14 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 25: Comparison: Control Group; Changes from post-test to Follow-up in the Relationship Quality subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.07, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 26: Comparison: Intervention; Changes from post-test to Follow-up in the Relationship Quality subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.05, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 27: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Relationship Quality subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.03, Standard Error of Mean 0.08 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 28: Comparison: Control Group; Changes from post-test to Follow-up in the Emotional Abuse subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.02, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 29: Comparison: Intervention; Changes from post-test to Follow-up in the Emotional Abuse subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — Changes from post-test to Follow-up in the Emotional Abuse subscale for the control group; Slope = 0, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 30: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Emotional Abuse subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.02, Standard Error of Mean 0.06 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 31: Comparison: Control Group; Changes from post-test to Follow-up in the Relationship Satisfaction subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0, Standard Error of Mean 0.01 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 32: Comparison: Intervention; Changes from post-test to Follow-up in the Relationship Satisfaction subscale for the interventionn group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.01, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 33: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Relationship satisfaction subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.01, Standard Error of Mean 0.02 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 34: Comparison: Control Group; Changes from post-test to Follow-up in the Relationship Commitment subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.03, Standard Error of Mean 0.02 — Changes from post-test to Follow-up in the Emotional Abuse subscale for the control group
Statistical Analysis 35: Comparison: Intervention; Changes from post-test to Follow-up in the Relationship Commitment subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.03, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 36: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Relationship Commitment subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.05, Standard Error of Mean 0.18 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 37: Comparison: Control Group; Change from pre-test to follow-up in banking subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.08, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 38: Comparison: Intervention; Change from pre-test to follow-up in banking subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.02, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 39: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in Banking subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.07, Standard Error of Mean 0.08 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 40: Comparison: Control Group; Change from post-test to follow-up in banking subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.11, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 41: Comparison: Intervention; Change from post-test to follow-up in banking subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.06, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 42: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in Banking subscale; Test type: Superiority; p < .10, Multilevel modeling — No adjustment to p value; Slope = -0.05, Standard Error of Mean 0.03; Changes from post-test to follow-up in the intervention group were not significantly different from the change from post-test to follow-up in the control group
Statistical Analysis 43: Comparison: Control Group; Change from pre-test to follow-up in Difficulty to Pay Bills for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.09, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 44: Comparison: Intervention; Change from pre-test to follow-up in Difficulties to Pay Bills subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.19, Standard Error of Mean 0.07 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 45: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in Difficulties to pay bills subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.1, Standard Error of Mean 0.09 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 46: Comparison: Control Group; Change from post-test to follow-up in Difficulty to Pay Bills subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 47: Comparison: Intervention; Change from post-test to follow-up in Difficulties to Pay Bills subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.02, Standard Error of Mean 0.03 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 48: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in Difficulty to Pay Bills subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.02, Standard Error of Mean 0.03 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 49: Comparison: Control Group; Change from pre-test to follow-up in depression subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p vallue; Slope = -0.69, Standard Error of Mean 0.21 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 50: Comparison: Intervention; Change from pre-test to follow-up in depression subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.72, Standard Error of Mean 0.25 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 51: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in Depression subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.03, Standard Error of Mean 0.32 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 52: Comparison: Control Group; Change from post-test to follow-up in depression subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.01, Standard Error of Mean 0.07 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 53: Comparison: Intervention; Change from post-test to follow-up in depression subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.09, Standard Error of Mean 0.07 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 54: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in depression subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.07, Standard Error of Mean 0.10 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 55: Comparison: Control Group; Change from pre-test to follow-up in the Anxiety subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.29, Standard Error of Mean 0.12; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 56: Comparison: Intervention; Change from pre-test to follow-up in the Anxiety subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.34, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 57: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in Anxiety subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.03, Standard Error of Mean 0.32 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 58: Comparison: Control Group; Change from post-test to follow-up in anxiety subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.03, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 59: Comparison: Intervention; Change from post-test to follow-up in anxiety subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.07, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 60: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in the Anxiety subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.1, Standard Error of Mean 0.06 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 61: Comparison: Control Group; Change from pre-test to follow-up in parenting stress subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.01, Standard Error of Mean 0.09 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 62: Comparison: Intervention; Change from pre-test to follow-up in parenting stress subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.09, Standard Error of Mean 0.1 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 63: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in parenting stress subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.1, Standard Error of Mean 0.13; Changes from pre-test to follow-up in the intervention group were not significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 64: Comparison: Control Group; Change from post-test to follow-up in banking subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.06, Standard Error of Mean 0.03 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 65: Comparison: Intervention; Change from post-test to follow-up in parenting stress subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.01, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 66: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in Parenting Stress subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.05, Standard Error of Mean 0.04 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 67: Comparison: Control Group; Change from pre-test to follow-up in Time with Partner subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling — No adjustment to p value; Slope = 0.26, Standard Error of Mean 0.13 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 68: Comparison: Intervention; Change from pre-test to follow-up in Time with Parter subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.22, Standard Error of Mean 0.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 69: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up inn Time with Partner subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.04, Standard Error of Mean 0.20 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 70: Comparison: Control Group; Change from post-test to follow-up in Time with Partner subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.14, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 71: Comparison: Intervention; Change from post-test to follow-up in Time with Partner subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.05, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 72: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in Time with Partner subscale; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.2, Standard Error of Mean 0.06; Changes from post-test to follow-up in the intervention group were significantly different from the change from post-test to follow-up in the control group
Statistical Analysis 73: Comparison: Control Group; Change from pre-test to follow-up in Conflict Management Satisfaction subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = 0.13, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 74: Comparison: Intervention; Change from pre-test to follow-up in Conflict Management Satisfaction subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = 0.32, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 75: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in Conflict Management Satisfaction subscale; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = 0.19, Standard Error of Mean 0.08 — Changes from pre-test to follow-up in the intervention group were significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 76: Comparison: Control Group; Change from post-test to follow-up in Conflict Management Satisfaction subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.01, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 77: Comparison: Intervention; Change from post-test to follow-up in conflict management satisfaction subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 78: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in Conflict Management Satisfaction subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0, Standard Error of Mean 0.02; [other analysis details as in outcome 3, analysis 42]
Statistical Analysis 79: Comparison: Control Group; Change from pre-test to follow-up in budgeting subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.1, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 80: Comparison: Intervention; Change from pre-test to follow-up in Budgeting subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.12, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 81: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up in Budgeting subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.22, Standard Error of Mean 0.07; Changes from pre-test to follow-up in the intervention group were significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 82: Comparison: Control Group; Change from post-test to follow-up in budgeting subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0., Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 83: Comparison: Intervention; Change from post-test to follow-up in budgeting subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.11, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 84: Comparison: Control Group vs Intervention; [analysis description as in outcome 3, analysis 81]; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = -0.1, Standard Error of Mean 0.02; [other analysis details as in outcome 3, analysis 81]

4. Primary Outcome: Brief Coping Orientation to Problems Experienced (COPE) Inventory- Baseline/Pre-test (Time1)
Description: The Brief Coping Orientation to Problems Experienced (COPE) Inventory was developed by Carver (1997)This is a 28 item self-report instrument that measures the respondent's individual coping strategies. The measure has 14 subscales: Self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Each subscale has two items. Only totals for each subscale are computed. Total subscale range: 0-6 for each. Higher scores represent more use of the particular coping strategy.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Baseline/Pre-test (Time 1) (Completed in first workshop session for Intervention Group and int the Intake and Enrollment Meeting for the Control Group)
Population: 294 individuals (147 couples) were assigned to control group but only 268 individuals (134 couples) completed the pre-test survey.
  290 individuals (145 couples) were assigned to the intervention group but only 212 individuals (106 couples) completed the pre-test survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Acceptance | 3.27 (1.73) | 3.45 (1.63)
  Active Coping | 4 (1.76) | 3.84 (1.6)
  Behavioral Disengagement | 0.52 (0.84) | 0.78 (0.86)
  Denial | 0.85 (1.38) | 0.89 (1.26)
  Humor | 1.62 (1.77) | 1.71 (1.71)
  Planning | 4.05 (1.77) | 4.02 (1.65)
  Positive Reframing | 3.24 (1.85) | 3.34 (1.76)
  Self-Blame | 2.41 (1.85) | 2.56 (1.83)
  Self-Distraction | 2.67 (1.76) | 3.21 (1.79)
  Substance Use | 0.62 (1.27) | 0.77 (1.41)
  Using Emotional Support | 2.31 (1.93) | 2.5 (2.08)
  Using Instrumental Support | 2.64 (1.94) | 2.71 (2.02)
  Venting | 2.26 (1.67) | 2.61 (1.55)

5. Primary Outcome: Brief Coping Orientation to Problems Experienced (COPE) Inventory - Post- Test (Time2)
Description: The Brief Coping Orientation to Problems Experienced (COPE) Inventory was developed by Carver (1997).This is a 28 item self-report instrument that measures the respondent's individual coping strategies. The measure has 14 subscales: Self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Each subscale has two items. Only totals for each subscale are computed. Total subscale range: 0-6 for each. Higher scores represent more use of the particular coping strategy.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: 294 individuals (147 couples) were assigned to control group but only 186 individuals (93 couples) completed the pre-test survey.
  290 individuals (145 couples) were assigned to the intervention group but only 144 individuals (72 couples) completed the pre-test survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Acceptance | 2.97 (1.86) | 3.62 (1.62)
  Active Coping | 3.55 (1.9) | 4.11 (1.78)
  Behavioral Disengagement | 0.54 (0.85) | 0.52 (0.86)
  Denial | 0.91 (1.46) | 0.63 (1.08)
  Humor | 1.77 (1.85) | 1.63 (1.69)
  Planning | 3.61 (1.87) | 4.38 (1.71)
  Positive Reframing | 2.99 (1.94) | 3.24 (1.82)
  Self-Blame | 1.81 (1.83) | 2.01 (1.67)
  Self-Distraction | 2.63 (1.72) | 2.65 (1.8)
  Substance Use | 0.76 (1.45) | 0.58 (1.26)
  Using Emotional Support | 2.22 (1.9) | 2.38 (1.91)
  Using Instrumental Support | 2.51 (1.98) | 2.71 (1.99)
  Venting | 1.93 (1.61) | 2.33 (1.58)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to posttest in the Acceptance subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling; Slope = -0.35, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to posttest in the Acceptance subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.33, Standard Error of Mean 0.14 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Acceptance subscale; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.68, Standard Error of Mean 0.18 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 4: Comparison: Control Group; Changes from pre-test to posttest in the Active Coping subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling; Slope = -0.34, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Changes from pre-test to posttest in the Active Coping subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.38, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Active Coping subscale; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.72, Standard Error of Mean 0.18; [other analysis details as in outcome 2, analysis 9]
Statistical Analysis 7: Comparison: Control Group; Changes from pre-test to posttest in the Planning subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling; Slope = -0.32, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Changes from pre-test to posttest in the Planning subscale for the intervention group; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.44, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Planning subscale; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.76, Standard Error of Mean 0.18 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 10: Comparison: Control Group; Changes from pre-test to posttest in the Instrumental Support subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.15, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Changes from pre-test to posttest in the Instrumental Support subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.03, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Instrumental Support subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.12, Standard Error of Mean 0.18 — [estimate comment as in outcome 2, analysis 21]

6. Primary Outcome: Brief Coping Orientation to Problems Experienced (COPE) Inventory - Six-month Follow-up (Time 3)
Description: as for outcome 5
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Acceptance | 2.71 (1.77) | 3.49 (1.51)
  Active Coping | 3.54 (1.86) | 4.17 (1.5)
  Behavioral Disengagement | 0.57 (0.92) | 0.6 (0.85)
  Denial | 0.93 (1.57) | 0.65 (1.14)
  Humor | 1.42 (1.69) | 1.47 (1.62)
  Planning | 3.55 (1.88) | 4.03 (1.75)
  Positive Reframing | 3.1 (1.93) | 3.22 (1.66)
  Self-Blame | 1.7 (1.76) | 2.26 (1.82)
  Self-Distraction | 2.34 (1.85) | 2.93 (1.51)
  Substance Use | 0.62 (1.38) | 0.69 (1.34)
  Using Emotional Support | 2 (1.77) | 2.7 (1.7)
  Using Instrumental Support | 2.39 (1.77) | 2.8 (1.67)
  Venting | 1.86 (1.67) | 2.21 (1.51)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to Follow-up in the Acceptance subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -0.36, Standard Error of Mean 0.14 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to Follow-up in the Acceptance subscale for the intervention group; Test type: Superiority; p < .05, Wilcoxon (Mann-Whitney); Slope = 0.41, Standard Error of Mean 0.18 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Aceptance subscale; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.77, Standard Error of Mean 0.22 — [estimate comment as in outcome 3, analysis 15]
Statistical Analysis 4: Comparison: Control Group; Changes from pre-test to Follow-up in the Active Coping subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -0.36, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Changes from pre-test to Follow-up in the Active Coping subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.40, Standard Error of Mean 0.18 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Active Coping subscale; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.76, Standard Error of Mean 0.22 — [estimate comment as in outcome 3, analysis 15]
Statistical Analysis 7: Comparison: Control Group; Changes from pre-test to Follow-up in the Planning subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -0.34, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Changes from pre-test to Follow-up in the Planning subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.59, Standard Error of Mean 0.18 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Planning subscale; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.94, Standard Error of Mean 0.23 — [estimate comment as in outcome 3, analysis 15]
Statistical Analysis 10: Comparison: Control Group; Changes from pre-test to Follow-up in the Instrumental Support subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.11, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Changes from pre-test to Follow-up in the Instrumental Support subscale for the Intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.02, Standard Error of Mean 0.18 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Instrumental Support subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.13, Standard Error of Mean 0.23 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 13: Comparison: Control Group; Changes from post-test to Follow-up in the Acceptance subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.02, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 14: Comparison: Intervention; Changes from post-test to Follow-up in the Acceptance subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.07, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 15: Comparison: Control Group vs Intervention; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.09, Standard Error of Mean 0.07 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 16: Comparison: Control Group; Test type: Superiority — Changes from post-test to Follow-up in the Active Coping subscale for the control group; p > .05, Multilevel modeling; Slope = 0.02, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 17: Comparison: Intervention; Changes from post-test to Follow-up in the Active Coping subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.03, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 18: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Active Copinng subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.04, Standard Error of Mean 0.07 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 19: Comparison: Control Group; Changes from post-test to Follow-up in the Plannning subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.02, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 20: Comparison: Intervention; Changes from post-test to Follow-up in the Planning subscale for the intervention group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -0.15, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 21: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Planning subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.17, Standard Error of Mean 0.07 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 22: Comparison: Control Group; Changes from post-test to Follow-up in the Instrumental Support subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.04, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 23: Comparison: Intervention; Changes from post-test to Follow-up in the Instrumental Support subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.05, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 24: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Instrumental Support subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.01, Standard Error of Mean 0.07 — [estimate comment as in outcome 3, analysis 21]

7. Primary Outcome: Brief Coping Orientation to Problems Experienced (COPE) Inventory in Relation to Financial Problems - Baseline/Pre-test (Time1)
Description: The Brief Coping Orientation to Problems Experienced (COPE) Inventory was developed by Carver (1997).This is a 28 item self-report instrument that measures the respondent's individual coping strategies. We have repeated the same 28 items but respondents had to answer about coping strategies in relationship to coping with financial issues in particular. The measure has 14 subscales: Self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Each subscale has two items. Only totals for each subscale are computed. Total subscale range: 0-6 for each. Higher scores represent more use of the particular coping strategy.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Acceptance | 3.25 (1.91) | 3.3 (1.64)
  Active Coping | 3.93 (1.79) | 3.93 (1.78)
  Behavioral Disengagement | 0.46 (0.83) | 0.54 (0.91)
  Denial | 0.9 (1.53) | 0.79 (1.26)
  Humor | 0.23 (1.68) | 1.01 (1.45)
  Planning | 4.13 (1.83) | 4 (1.8)
  Positive Reframing | 2.89 (1.93) | 2.78 (1.9)
  Self-Blame | 2.19 (2.09) | 2.32 (1.97)
  Self-Distraction | 2.24 (1.8) | 2.47 (1.86)
  Substance Use | 0.46 (1.14) | 0.63 (1.31)
  Using Emotional Support | 1.85 (1.92) | 1.8 (1.76)
  Using Instrumental Support | 2.34 (1.95) | 2.25 (1.79)
  Venting | 1.99 (1.7) | 2.13 (1.61)

8. Primary Outcome: Brief Coping Orientation to Problems Experienced (COPE) Inventory in Relation to Financial Problems - Post- Test (Time2)
Description: The Brief Coping Orientation to Problems Experienced (COPE) Inventory was developed by Carver (1997). This is a 28 item self-report instrument that measures the respondent's individual coping strategies. We have repeated the same 28 items but respondents had to answer about coping strategies in relationship to coping with financial issues in particular. The measure has 14 subscales: Self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Each subscale has two items. Only totals for each subscale are computed. Total subscale range: 0-6 for each. Higher scores represent more use of the particular coping strategy.
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Acceptance | 2.99 (1.84) | 3.73 (1.67)
  Active Coping | 3.65 (1.91) | 4.2 (1.79)
  Behavioral Disengagement | 0.57 (0.91) | 0.35 (0.78)
  Denial | 0.97 (1.55) | 0.47 (1.04)
  Humor | 1.42 (1.7) | 1.36 (1.58)
  Planning | 3.61 (1.99) | 4.35 (1.77)
  Positive Reframing | 2.73 (1.96) | 3.02 (1.77)
  Self-Blame | 1.85 (1.93) | 1.74 (1.67)
  Self-Distraction | 2.17 (1.81) | 2.31 (1.73)
  Substance Use | 0.63 (1.37) | 0.43 (1.03)
  Using Emotional Support | 1.94 (1.92) | 2.18 (1.87)
  Using Instrumental Support | 2.28 (1.96) | 2.87 (2.04)
  Venting | 1.75 (1.62) | 2.07 (1.51)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to posttest in the Acceptance subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling; Slope = -0.3, Standard Error of Mean 0.12 — Changes from pre-test to Follow-up in the Emotional Abuse subscale for the control group
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to posttest in the Emotional Abuse subscale for the control group; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.47, Standard Error of Mean 0.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.77, Standard Error of Mean 0.19 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 4: Comparison: Control Group; Changes from pre-test to posttest in the Active Coping subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.17, Standard Error of Mean 0.13 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Changes from pre-test to posttest in the Active Coping subscale for the intervention group; Test type: Superiority; p < .10, Multilevel modeling; Slope = 0.30, Standard Error of Mean 0.17 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.47, Standard Error of Mean 0.2 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 7: Comparison: Control Group; Changes from pre-test to posttest in the Planning subscale for the control group; Test type: Superiority; p < .05, Multilevel modeling; Slope = -0.38, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Changes from pre-test to posttest in the Planning subscale for the Intervention group; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.37, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p < .001, Multilevel modeling; Slope = 0.74, Standard Error of Mean 0.19 — [estimate comment as in outcome 2, analysis 14]
Statistical Analysis 10: Comparison: Control Group; Changes from pre-test to posttest in the Instrumental Support subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.11, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Changes from pre-test to posttest in the Instrumental Support subscale for the intervention group; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.49, Standard Error of Mean 0.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.60, Standard Error of Mean 0.19 — [estimate comment as in outcome 2, analysis 14]

9. Primary Outcome: Brief Coping Orientation to Problems Experienced (COPE) Inventory in Relation to Financial Problems - Six-month Follow-up (Time 3)
Description: as for outcome 8
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Acceptance | 2.78 (1.86) | 3.74 (1.66)
  Active Coping | 3.4 (1.95) | 4.11 (1.74)
  Behavioral Disengagement | 0.6 (1.01) | 0.49 (0.91)
  Denial | 0.9 (1.54) | 0.64 (1.19)
  Humor | 1.14 (1.58) | 1.13 (1.58)
  Planning | 3.41 (2.05) | 4.42 (1.68)
  Positive Reframing | 2.91 (2.07) | 2.69 (1.73)
  Self-Blame | 1.49 (1.72) | 2.26 (1.76)
  Self-Distraction | 1.92 (1.69) | 2.28 (1.56)
  Substance Use | 0.49 (1.18) | 0.54 (1.22)
  Using Emotional Support | 1.73 (1.86) | 2.29 (1.89)
  Using Instrumental Support | 2.04 (1.84) | 2.54 (1.78)
  Venting | 1.51 (1.62) | 1.94 (1.44)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to Follow-up in the Acceptance subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.25, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to Follow-up in the Acceptance subscale for the intervention group; Test type: Superiority; p < .01, Multilevel modeling; Slope = .52, Standard Error of Mean 0.19 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up in the Acceptance subscale; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.78, Standard Error of Mean 0.24; The expected increase from pre-test to follow-up in the intervention group is significantly different from the change from pre-test to follow-up in the control group
Statistical Analysis 4: Comparison: Control Group; Changes from pre-test to Follow-up in the Active Coping subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.09, Standard Error of Mean 0.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Changes from pre-test to Follow-up in the Active Coping subscale for the intervention group; Test type: Superiority; p < .10, Multilevel modeling; Slope = 0.36, Standard Error of Mean 0.2 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p < .10, Multilevel modeling; Slope = 0.40, Standard Error of Mean 0.25 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 7: Comparison: Control Group; Changes from pre-test to Follow-up in the Planning subscale for the control group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -0.31, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Changes from pre-test to Follow-up in the Planning subscale for the intervention group; Test type: Superiority; p < .05, Multilevel modeling; Slope = 0.40, Standard Error of Mean 0.18 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.71, Standard Error of Mean 0.23 — [estimate comment as in outcome 3, analysis 15]
Statistical Analysis 10: Comparison: Control Group; Changes from pre-test to Follow-up in the Instrumental Support subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.02, Standard Error of Mean 0.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Changes from pre-test to Follow-up in the Instrumental Support subscale for the intervention group; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.64, Standard Error of Mean 0.19 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; [analysis description as in outcome 6, analysis 12]; Test type: Superiority; p < .01, Multilevel modeling; Slope = 0.66, Standard Error of Mean 0.24 — [estimate comment as in outcome 3, analysis 15]
Statistical Analysis 13: Comparison: Control Group; Changes from post-test to Follow-up in the Acceptance subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.05, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 14: Comparison: Intervention; Changes from post-test to Follow-up in the Acceptance subscale for the interventionn group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.06, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 15: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Acceptance subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.01, Standard Error of Mean 0.08 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 16: Comparison: Control Group; Changes from post-test to Follow-up in the Active Coping subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.08, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 17: Comparison: Intervention; Changes from post-test to Follow-up in the Active Coping in the intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.07, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 18: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Active Coping subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.01, Standard Error of Mean 0.08 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 19: Comparison: Control Group; Changes from post-test to Follow-up in the Planning subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.07, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 20: Comparison: Intervention; Changes from post-test to Follow-up in the Planning subscale for the intervention group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.04, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 21: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in Planning subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.03, Standard Error of Mean 0.07 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 22: Comparison: Control Group; Changes from post-test to Follow-up in the Instrumental Support subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.09, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 23: Comparison: Intervention; Changes from post-test to Follow-up in the Instrumental Support subscale for the intervention group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -0.15, Standard Error of Mean 0.06 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 24: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up in the Instrumental Supportt subscale; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.06, Standard Error of Mean 0.08 — [estimate comment as in outcome 3, analysis 21]

10. Primary Outcome: Family Economic Strain Scale - Baseline/Pre-test (Time 1)
Description: Developed by Hilton and Devall (1997). This is a 15-item self-report instrument that measures the respondent's level of economic strain.As not all couples had children, the two items related to children were excluded. Scale range: 13-65. Higher scores represent higher economic strain
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale | 29.02 (27.52) | 30.98 (11.02)

11. Primary Outcome: Family Economic Strain Scale - Post-test (Time 2)
Description: as for outcome 10
Time Frame: Post-test (8weeks after pre-test/Time1)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale | 27.52 (10) | 30.35 (10.65)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to posttest for the control group; Test type: Superiority; p < .05, Multilevel modeling; Slope = -1.41, Standard Error of Mean 0.49; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to posttest for the intervention group; Test type: Superiority; p < .01, Multilevel modeling; Slope = 2.02, Standard Error of Mean 0.69 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.62, Standard Error of Mean 0.83 — Changes from pre-test to post-test t in the intervention group were not significantly different from the change from pre-test to post-test in the control group

12. Primary Outcome: Family Economic Strain Scale - Six-month Follow-up (Time 3)
Description: as for outcome 10
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale | 26.44 (10.36) | 27.33 (8.61)
Statistical Analysis 1: Comparison: Control Group; Changes from pre-test to Follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -1.48, Standard Error of Mean 0.6 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Changes from pre-test to Follow-up for the intervention group; Test type: Superiority; p < .10, Multilevel modeling; Slope = -1.5, Standard Error of Mean 0.82 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Follow-up; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.02, Standard Error of Mean 1.01 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 4: Comparison: Control Group; Changes from post-test to Follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = 0.08, Standard Error of Mean 0.02 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Changes from post-test to Follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.52, Standard Error of Mean 0.23 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Post-test to Follow-up; Test type: Superiority; p > .05, Multilevel modeling; Slope = -0.6, Standard Error of Mean 0.03 — [estimate comment as in outcome 3, analysis 21]

13. Primary Outcome: Difficulties in Emotion Regulation - Baseline/Pre-test (Time 1)
Description: Developed by Gratz and Roemer (2004). This is a 36-item self-report instrument that measures the respondent difficulties in emotion regulation. Scale range: 36-180. Higher scores represent more difficulties in emotion regulation
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale | 70.78 (19.91) | 78.85 (22.43)

14. Primary Outcome: Difficulties in Emotion Regulation - Post-test (Time 2)
Description: as for outcome 13
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale | 72.95 (20.5) | 75.58 (19.54)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to post-test in Difficulties in Emotion Regulation for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment for p value; Slope = -0.34, Standard Error of Mean 1.16 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to post-test for the intervention group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment for p value; Slope = -3.07, Standard Error of Mean 1.51 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -2.74, Standard Error of Mean 1.85 — [estimate comment as in outcome 2, analysis 39]

15. Primary Outcome: Difficulties in Emotion Regulation - Six-month Follow-up (Time 3)
Description: as for outcome 13
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale | 70.32 (22.76) | 74.92 (20.22)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.7, Standard Error of Mean 1.41; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -2.74, Standard Error of Mean 1.79 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -2.04, Standard Error of Mean 2.24 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 4: Comparison: Control Group; Change from post-test to follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = 0.36, Standard Error of Mean 0.46 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from post-test to follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.33, Standard Error of Mean 0.5 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.69, Standard Error of Mean 0.68 — [estimate comment as in outcome 3, analysis 21]

16. Primary Outcome: Conflict Tactics Scales-R - Baseline/Pre-test (Time 1)
Description: Developed by Straus, Comby, Boney-McCoy, & Sugarman (1996). This 78-item self report instrument measures physical assault (12 items), physical injury (6 items), psychological aggression (8 items), sexual coercion (7 items) and negotiation (6 items) by the respondent and by the partner. Only the physical assault and psychological aggression subscales were considered for analysis in this study. A total prevalence score for each subscale was calculated. Total prevalence scores ranged 0 to 12 for the physical assault subscale and from 0 to 8 for the psychological aggresion subscale. Higher total scores represented higher levels of the variable. For the psychological aggression and physical assault subscales only the partner with the higher score was considered due to underreporting of these behaviors.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Psychological Aggression | 2.06 (1.73) | 2.36 (1.7)
  Physical Assault | 0.37 (1.12) | 0.38 (0.97)

17. Primary Outcome: Conflict Tactics Scales-R Post-test (Time 2)
Description: as for outcome 16
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Psychological Aggression | 1.54 (1.68) | 1.54 (1.58)
  Physical Assault | 0.5 (1.87) | 0.11 (0.51)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to post-test in psychological agggression subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.39, Standard Error of Mean 0.11 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to post-test in psychological aggression subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.73, Standard Error of Mean 0.14 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Psychological Aggression subscale; Test type: Superiority; p < .10, Multilevel modeling — No adjustment to p value; Slope = -0.34, Standard Error of Mean 0.17 — [estimate comment as in outcome 2, analysis 39]
Statistical Analysis 4: Comparison: Control Group; Change from pre-test to post-test in physical assault subscale for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0, Standard Error of Mean 0.09; A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from pre-test to post-test in the physical assault subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.34, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Physical Assault subscale; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.34, Standard Error of Mean 0.14 — Changes from pre-test to post-test in the intervention group were significantly different from the change from pre-test to pos-test in the control group

18. Primary Outcome: Conflict Tactics Scales-R - Six Month Follow-up (Time 3)
Description: as for outcome 16
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Psychological Aggression | 1.94 (2.08) | 1.85 (1.96)
  Physical Assault | 0.58 (2.11) | 0.38 (1.81)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to follow-up in the psychological aggression subscale for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.47, Standard Error of Mean 0.13 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to follow-up in the Psychological Aggression subscale for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -0.77, Standard Error of Mean 0.17 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up inn the psychological aggression subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.30, Standard Error of Mean 0.21 — [estimate comment as in outcome 2, analysis 27]
Statistical Analysis 4: Comparison: Control Group; Change from post-test to follow-up for the control group in the psychological aggression subscale; Test type: Superiority; p < .10, Multilevel modeling — No adjustment to p value; Slope = 0.08, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from post-test to follow-up for the intervention group for the psychological aggresssion subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.04, Standard Error of Mean 0.05 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up in the psychological aggression subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.04, Standard Error of Mean 0.06 — [estimate comment as in outcome 3, analysis 21]
Statistical Analysis 7: Comparison: Control Group; Change from pre-test to follow-up for the control group for the physical assault subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.03, Standard Error of Mean 0.12 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Change from pre-test to follow-up for the control group for the Physical Assault Subscale; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.40, Standard Error of Mean 0.15 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up for the Physical Assault subscale; Test type: Superiority; p < .05, Multilevel modeling — No adjustment to p value; Slope = -0.37, Standard Error of Mean 0.18 — [estimate comment as in outcome 3, analysis 75]
Statistical Analysis 10: Comparison: Control Group; Change from post-test to follow-up for the control group for the Physical Assault subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.02, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 11: Comparison: Intervention; Change from post-test to follow-up for the intervention group for the Physical Assault subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.06, Standard Error of Mean 0.04 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 12: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.04, Standard Error of Mean 0.06 — [estimate comment as in outcome 3, analysis 21]

19. Primary Outcome: Depression, Anxiety, and Stress Scale - Stress Subscale Baseline/Pre-test (Time 1)
Description: Developed by Lovibond & Lovibond (1995). The stress subscale has 7 items and scale range is 0-21. Higher scores represent more symptoms of stress
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale | 13.47 (10.01) | 17.14 (8.45)

20. Primary Outcome: Depression, Anxiety, and Stress Scale - Stress Subscale Post-test (Time 2)
Description: as for outcome 19
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale | 11.87 (10.13) | 11.88 (8.85)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to post-test for the control group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment to p value; Slope = -2.12, Standard Error of Mean 0.57 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to post-test for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment in p value; Slope = -4.46, Standard Error of Mean 0.73 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in Time; Test type: Superiority; p < .05, Multilevel modeling — No adjustment in p value; Slope = -2.34, Standard Error of Mean 0.89 — [estimate comment as in outcome 17, analysis 6]

21. Primary Outcome: Depression, Anxiety, and Stress Scale - Stress Subscale Six-month Follow up (Time 3)
Description: as for outcome 19
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale | 10.44 (8.54) | 12.77 (7.79)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to follow-up for the control group; Test type: Superiority; p < .05, Multilevel modeling — No adjustment in p value; Slope = -1.96, Standard Error of Mean 0.7 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to follow-up for the intervention group; Test type: Superiority; p < .001, Multilevel modeling — No adjustment in p value; Slope = -4.48, Standard Error of Mean 0.88 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up; Test type: Superiority; p < .05, Multilevel modeling — No adjustment in p value; Slope = -2.52, Standard Error of Mean 1.1 — [estimate comment as in outcome 3, analysis 75]
Statistical Analysis 4: Comparison: Control Group; Change from post-test to follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = -0.16, Standard Error of Mean 0.24 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from post-test to follow-up for the control group; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.03, Standard Error of Mean 0.26 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from post-test to follow-up; Test type: Superiority; p > .05, Multilevel modeling — No adjustment to p value; Slope = 0.19, Standard Error of Mean 0.35 — [estimate comment as in outcome 3, analysis 21]

22. Primary Outcome: Dyadic Coping Inventory - Baseline/Pre-test (Time 1)
Description: Developed by Guy Bodenmann (2008). This 37-item self-report instrument measures how couples cope with stress in general. It includes stress communication, supportive dyadic coping, delegated dyadic coping, common dyadic coping, negative dyadic coping, and evaluation of dyadic coping. Only the communication (4 items by self and 4 items by partner), supportive (5 items by self and 5 items by partner), negative (4 items by self and 4 items by partners), and common dyadic coping (5 items) subscales were used in the present study. Response options range from 1 to 5 . Total scores for each subscale were computed. Subscale total scores ranged from 4 to 20 for Stress Communication, 5 to 25 for Supportive, 4 to 20 for Negative, and 5 to 25 for Common Dyadic Coping. Higher scores mean higher frequency of use of that coping behaviors.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Common Dyadic Coping | 16.75 (5.26) | 15.96 (4.63)
  Supportive Dyadic Coping | 18.29 (3.93) | 17.83 (3.35)
  Negative Dyadic Coping | 17.76 (6.75) | 17.75 (5.42)
  Stress Communication | 14.06 (2.93) | 13.84 (2.41)

23. Primary Outcome: Dyadic Coping Inventory - Post-Test (Time 2)
Description: as for outcome 22
Time Frame: Post-test: 8 weeks after Pre-Test ; Follow-up: 6 months after Post-Test
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Common Dyadic Coping | 17.26 (5.41) | 16.84 (4.57)
  Supportive Dyadic Coping | 18.37 (4.02) | 18.46 (3.17)
  Negative Dyadic Coping | 16.97 (7.13) | 16.74 (6.07)
  Stress Communication | 14.38 (2.86) | 14.25 (2.45)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to post-test for the control group for Supportive Dyadic Coping subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.37, Standard Error of Mean 0.24 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to post-test for the intervention group; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.71, Standard Error of Mean 0.31 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test in the Supportive Dyadic Coping subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.33, Standard Error of Mean 0.38; [other analysis details as in outcome 2, analysis 30]
Statistical Analysis 4: Comparison: Control Group; Change from pre-test to post-test for the control group for the common dyadic coping subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.23, Standard Error of Mean 0.3 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from pre-test to post-test for the intervention group in the Common Dyadic Coping subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.21, Standard Error of Mean 0.39 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test for the Common Dyadic Coping Subscale; Test type: Superiority; p < .10, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.97, Standard Error of Mean 0.47 — [estimate comment as in outcome 2, analysis 21]
Statistical Analysis 7: Comparison: Control Group; Change from pre-test to post-test for the control group in the Negative Dyadic Coping Subscale; Test type: Superiority; p < .10, Multilevel modeling — No adjustment in p value; Slope = -0.74, Standard Error of Mean 0.37 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Change from pre-test to post-test for the intervention group for the Negative Dyadic Coping subscale; Test type: Superiority; p < .05, Multilevel modeling — No adjustment in p value; Slope = -1.14, Standard Error of Mean 0.49 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test inn the Negative Dyadic Coping Scale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.39, Standard Error of Mean 0.60 — [estimate comment as in outcome 2, analysis 21]

24. Primary Outcome: Dyadic Coping Inventory - Follow-up (Time 3)
Description: as for outcome 22
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Common Dyadic Coping | 17.51 (5.55) | 17.29 (4.55)
  Supportive Dyadic Coping | 18.22 (4.61) | 18.61 (3.3)
  Negative Dyadic Coping | 15.91 (6.17) | 15.83 (5.83)
  Stress Communication | 13.71 (3.00) | 13.99 (2.69)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to follow-up for the control group for the Supportive Dyadic Coping Subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.57, Standard Error of Mean 0.29 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to follow-up for the intervention group for the Supportive Dyadic Coping Subscale; Test type: Superiority; p < .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.7, Standard Error of Mean 0.37 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from pre-test to follow-up for the Supportive Dyadic Coping Subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.19, Standard Error of Mean 0.46 — [estimate comment as in outcome 2, analysis 27]

25. Primary Outcome: Dyadic Coping With Economic Stress Inventory - Baseline/Pre-Test (Time 1)
Description: 34-item self-report instrument adapted from the Dyadic Coping Inventory to describe coping with economic stress. It includes stress communication, supportive dyadic coping, delegated dyadic coping, common dyadic coping, negative dyadic coping, and evaluation of dyadic coping. Only the communication (2 items by self and 2 items by partner), supportive (5 items by self and 5 items by partner), negative (4 items by self and 4 items by partners), and common dyadic coping (5 items) subscales were used in the present study. Response options range from 1 to 5. A total was caculated for each subscale by adding all responses. The total score for stress communication ranged from 2 to 10, supportive from 5 to 25, negative from 4 to 20, and common dyadic coping from 5 to 25. Higher scores mean higher frequency of use of that coping behaviors.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Common Dyadic Coping | 16.43 (5.81) | 15.69 (5.18)
  Supportive Dyadic Coping | 17.54 (4.22) | 17.19 (3.66)
  Negative Dyadic Coping | 18.76 (6.82) | 18.97 (6.18)
  Stress Communication | 5.77 (1.78) | 5.84 (1.61)

26. Primary Outcome: Dyadic Coping With Economic Stress Inventory - Post-Test (Time 2)
Description: This 34-item self-report instrument is an adaptation of the Dyadic Coping Inventory to economic stress and measures how couples cope with economic stress. Only the communication (2 items by self and 2 items by partner), supportive (5 items by self and 5 items by partner), negative (4 items by self and 4 items by partners), and common dyadic coping (5 items) subscales were used in the present study. Response options range from 1 to 5. A total was caculated for each subscale by adding all responses. The total score for stress communication ranged from 2 to 10, supportive from 5 to 25, negative from 4 to 20, and common dyadic coping from 5 to 25. Higher scores mean higher frequency of use of that coping behaviors.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Common Dyadic Coping | 16.78 (5.84) | 17.46 (4.83)
  Supportive Dyadic Coping | 17.65 (4.49) | 18.43 (3.9)
  Negative Dyadic Coping | 17.99 (7.27) | 17.98 (6.52)
  Stress Communication | 5.63 (1.83) | 6.0 (1.64)
Statistical Analysis 1: Comparison: Control Group; Change from pre-test to post-test for the control group in the Supportive Dyadic Coping Subcale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.03, Standard Error of Mean 0.26 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 2: Comparison: Intervention; Change from pre-test to post-test for the intervention group in the Supportive Dyadic Coping Scale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.45, Standard Error of Mean 0.33 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 3: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.42, Standard Error of Mean 0.41 — Changes from pre-test to post-test in the intervention group were significantly different from the change from pre-test to post-test in the control group
Statistical Analysis 4: Comparison: Control Group; Change from pre-test to post-test for the control group for the Common Dyadic Coping Subscale; Test type: Superiority; p > .05, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 0.22, Standard Error of Mean 0.35 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 5: Comparison: Intervention; Change from pre-test to post-test for the intervention group in the Common Dyadic Coping Subscale; Test type: Superiority; p < .001, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 2.12, Standard Error of Mean 0.45 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 6: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test inn the Common Dyadic Coping subscale; Test type: Superiority; p < .01, Multilevel modeling — [p-value comment as in outcome 2, analysis 1]; Slope = 1.91, Standard Error of Mean 0.55 — [estimate comment as in outcome 26, analysis 3]
Statistical Analysis 7: Comparison: Control Group; Change from pre-test to post-test for the control group for the Negative Dyadic Coping Scale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.68, Standard Error of Mean 0.42 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 8: Comparison: Intervention; Change from pre-test to post-test for the intervention group for the Negative Dyadic Coping Scale; Test type: Superiority; p < .10, Multilevel modeling — No adjustment in p value; Slope = -1.02, Standard Error of Mean 0.53 — A positive value indicates an increase while a negative value indicates a decrease
Statistical Analysis 9: Comparison: Control Group vs Intervention; Difference between the control and the intervention group in the change from Pre-test to Post-test for the Negative Dyadic Coping Subscale; Test type: Superiority; p > .05, Multilevel modeling — No adjustment in p value; Slope = -0.34, Standard Error of Mean 0.65 — [estimate comment as in outcome 2, analysis 21]

27. Primary Outcome: Dyadic Coping With Economic Stress Inventory - Six-month Follow-up (Time 3)
Description: as for outcome 26
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Common Dyadic Coping | 16.58 (5.77) | 17.46 (4.83)
  Supportive Dyadic Coping | 17.41 (4.88) | 18.43 (3.9)
  Negative Dyadic Coping | 18.79 (6.82) | 17.98 (6.52)
  Stress Communication | 5.68 (1.52) | 5.85 (1.36)

28. Primary Outcome: The Brief Communication Patterns Questionnaire - General and In Relation to Money Problems - Pre-test (Time 1)
Description: This is an 11-item self-report questionnaire that assesses the couple's demand/withdraw communication patterns as well as their level of constructive communication when there is a problem. Each item is responded on a scale from 1 to 9. The Demand/Withdraw Total Scale has 6 items. and the total score for the subscale ranges from 6 to 54 . The constructive communication subscale includes 3 items and. the total score for the subscale ranges from 3 to 27. Higher scores represent more occurrence of the communication pattern.The same eleven items were asked about communication behaviors in relation to money problems and scored in the same way.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Pre-test (Time 1) (Completed in first workshop session for Intervention Group and int the Intake and Enrollment Meeting for the Control Group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Demand/Withdraw General | 24.43 (11.58) | 25.87 (10.74)
  Demand/Withdraw for Money | 21.35 (11.87) | 21.10 (11.51)
  Constructive. Communication General | 19.02 (6.15) | 18.67 (5.72)
  Constructive Communication for Money Issues | 18.59 (6.68) | 18.95 (6.07)

29. Primary Outcome: The Brief Communication Patterns Questionnaire - General and In Relation to Money Problems - Post-test (Time 2)
Description: Developed by Futris, Campbell, Nielsen, & Burwell (2010). This is an 11-item self-report questionnaire that assesses the couple's demand/withdraw communication patterns as well as their level of constructive communication when there is a problem. Each item is responded on a scale from 1 to 9. The Demand/Withdraw Total Scale has 6 items. and the total score for the subscale ranges from 6 to 54 . The constructive communciation subscale includes 3 items and. the total score for the subscale ranges from 3 to 27. Higher scores represent more occurrence of the communication pattern.The same eleven items were asked about communication behaviors in relation to money problems and scored in the same way.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Post-test (8weeks after pre-test/Time1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Demand/Withdraw General | 21.68 (10.66) | 21.21 (10.02)
  Demand/Withdraw for Money Issues | 18.86 (11.95) | 17.08 (9.83)
  Constructive Communication General | 18.91 (6.13) | 19.99 (5.39)
  Constructive Communication for Money Issues | 18.95 (6.65) | 20.54 (5.62)

30. Primary Outcome: The Brief Communication Patterns Questionnaire - General and In Relation to Money Problems - Six-month Follow-up (Time 3)
Description: as for outcome 29
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Demand/Withdraw General | 22.25 (10.01) | 24.89 (10.76)
  Demand/Withdraw for Money Issues | 19.66 (11.25) | 19.95 (9.49)
  Constructive Communication General | 20.11 (5.50) | 20.19 (5.21)
  Constructive Communication for Money Issues | 20.00 (6.20) | 19.43 (5.68)

31. Primary Outcome: Financial Self-Efficacy Scale - Pre-test (Time 1)
Description: Developed by Dietz, Carrozza & Ritchey (2011). This is a 3-item self-report questionnaire that assesses the respondent's financial self-efficacy. Scale range 4-12. Higher scores represent higher financial self-efficacy
Time Frame: Pre-test (Time1Pre-test (Time 1) (Completed in first workshop session for Intervention Group and int the Intake and Enrollment Meeting for the Control Group)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale | 9.1 (2.6) | 8.53 (2.37)

32. Primary Outcome: Financial Self-Efficacy Scale - Post-test (Time 2)
Description: as for outcome 31
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale | 9.47 (2.38) | 9.38 (2.51)

33. Primary Outcome: Financial Self-Efficacy Scale - Six-month Follow-up (Time 3)
Description: as for outcome 31
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale | 9.25 (2.63) | 9.12 (2.45)

34. Primary Outcome: Revised Financial Management Behavior Scale - Pre-test (Time 1)
Description: Developed by Dew and Xiao (2011). This is a 15-item self-report questionnaire that assesses the respondent's financial management behavior. It includes four subscales: Insurance (3 items; scale range: 3-15), Credit management (3 items; scale range: 3-15), Savings (3 items; scale range: 3-15), Cash management (4 items; scale range: 4-20). Higher scores for each of the subscale depict healthy financial management practices.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Cash Management | 13.55 (3.79) | 14.03 (3.31)
  Credit Management | 9.97 (2.98) | 9.87 (3.16)
  Insurance | 10.74 (4.04) | 10.26 (4.13)
  Savings and Investment | 12.86 (5.81) | 12.32 (5.22)

35. Primary Outcome: Revised Financial Management Behavior Scale - Post-test (Time 2)
Description: as for outcome 34
Time Frame: Post-test (8weeks after pre-test/Time1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Cash Management | 14.28 (3.62) | 14.72 (2.98)
  Credit Management | 10.03 (3.22) | 9.64 (3.27)
  Insurance | 11.35 (3.86) | 10.79 (3.95)
  Savings and Investment | 14.34 (5.67) | 13.36 (5.38)

36. Primary Outcome: Revised Financial Management Behavior Scale - Six-month Follow-up(Time 3)
Description: as for outcome 34
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Cash Management | 14.60 (3.72) | 15.12 (2.99)
  Credit Management | 10.46 (3.09) | 10.30 (3.03)
  Insurance | 11.49 (3.87) | 11.16 (3.51)
  Savings and Investment | 15.11 (5.90) | 14.14 (4.86)

37. Primary Outcome: Financial Services Survey From FINRA - Pre-test (Time 1)
Description: Developed by FINRA for the National Financial Capability Study. This is a 5-item self-report questionnaire that assesses the respondent's use of financial services. Examples of specific items included "Taken out an auto title loan," "Taken out a short term "payday" loan," and "Used a pawn shop.". The measurement used a 5-point scale, ranging from 1(never) to 5 (4 or more times). Scale ranges from 5-25. Higher sores represent higher use of non-banking borrowing/alternative borrowing methods.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale | 5.87 (2.24) | 5.67 (1.77)

38. Primary Outcome: Financial Services Survey From FINRA - Post-test (Time 2)
Description: Developed by FINRA for the National Financial Capability Study. This is a 5-item self-report questionnaire that assesses the respondent's use of financial services. Examples of specific items included "Taken out an auto title loan," "Taken out a short term "payday" loan," and "Used a pawn shop.". The measurement used a 5-point scale, ranging from 1 (never) to 5 (4 or more times). Scale ranges from 5-25. Higher sores represent higher use of non-banking borrowing/alternative borrowing methods.
Time Frame: Post-test (8weeks after pre-test/Time1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale | 5.51 (1.62) | 5.61 (1.98)

39. Primary Outcome: Financial Services Survey From FINRA - Six-month Follow-up (Time 3)
Description: Developed by FINRA for the National Financial Capability Study. This is a 5-item self-report questionnaire that assesses the respondent's use of financial services. Examples of specific items included "Taken out an auto title loan," "Taken out a short term "payday" loan," and "Used a pawn shop.". The measurement used a 5-point scale, ranging from 1 (never) to 5 (4 or more times). Scale ranges from 5-25. Higher sores represent higher use of non-banking borrowing/alternative borrowing methods.
  The PI and data for this study are no longer available for query. There is no additional information at this time.
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale | 5.77 (2.45) | 5.40 (1.68)

40. Primary Outcome: Shared Goals and Values - Pre-test (Time 1)
Description: Developed by Archuleta, Grable, & Britt (2010) . This is a 4-item self-report questionnaire that assesses the respondent's perception of the extent to which he or she share financial goals and values with his/her partner. Scale range: 4-28. Higher scores represent more sharing
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale | 18.94 (6.97) | 20.41 (6.09)

41. Primary Outcome: Shared Goals and Values - Post-test (Time 2)
Description: Developed by Archuleta, Grable, & Britt (2010) .This is a 4-item self-report questionnaire that assesses the respondent's perception of the extent to which he or she share financial goals and values with his/her partner. Scale range: 4-28. Higher scores represent more sharing
Time Frame: Post-test (8weeks after pre-test/Time1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale | 20.64 (6.69) | 22.25 (5.3)

42. Primary Outcome: Shared Goals and Values - Six-month Follow-up (Time 3)
Description: as for outcome 41
Time Frame: Six-month follow up (six months after post-test/Time2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale | 19.18 (7.53) | 21.58 (5.49)

43. Primary Outcome: Couple Financial Management Roles and Satisfaction - Pre-Test (Time 1)
Description: There are two different 7-point Likert-type scales used for Financial Management Roles (FMR). The first part assesses spousal involvement in specific financial management roles. The scale ranges from 1 (FMR was primarily the participant's responsibility) to 7 (FMR was the spouse's primary responsibility). Scores were recoded (1 recoded to -3; 4 recoded to 0; and 7 recoded to 3). Scale ranges from -39 to 39. Lower score indicates the participant is more responsible and higher score the participant is less responsible for the FMR in his/her household. Second part of the FMR assesses respondents' level of satisfaction of their involvement in financial roles. The scale ranges from 1 (participant unsatisfied in his/her involvement) to 7 (participant satisfied in his/her involvement). Higher score indicates participant's satisfaction of involvement in specific financial role. Scale ranges from 13 to 91. The PI and data for this study are no longer available for query.
Time Frame: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  FMR Involvement | -0.59 (1.30) | -0.51 (1.39)
  FMR Participation | 6.88 (3.91) | 7.18 (3.50)

44. Primary Outcome: Couple Financial Management Roles and Satisfaction - Post-Test (Time 2)
Description: Developed by Archuleta (2008). This is a 13-item self-report questionnaire. There are two different 7-point Likert-type scales used for Financial Management Roles (FMR). The first part assesses spousal involvement in specific financial management roles. The scale ranges from 1 (FMR was primarily the participant's responsibility) to 7 (FMR was the spouse's primary responsibility). Scores were recoded (1 recoded to -3; 4 recoded to 0; and 7 recoded to 3). Scale ranges from -39 to 39. Lower score indicates the participant is more responsible and higher score the participant is less responsible for the FMR in his/her household. Second part of the FMR assesses respondents' level of satisfaction of their involvement in financial roles. The scale ranges from 1 (participant unsatisfied in his/her involvement) to 7 (participant satisfied in his/her involvement). Higher score indicates participant's satisfaction of involvement in specific financial role. Scale ranges from 13 to 91.
Time Frame: Post-test (8weeks after pre-test/Time1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  FMR Involvement | -0.44 (1.28) | -0.43 (1.29)
  FMR Participation | 7.73 (4.22) | 8.19 (3.77)

45. Primary Outcome: Couple Financial Management Roles and Satisfaction - Six-month Follow-up (Time 3)
Description: as for outcome 44
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  FMR Involvement | -0.77 (1.36) | -0.48 (1.33)
  FRM Participation | 7.78 (3.91) | 9.83 (2.48)

46. Primary Outcome: Perceived Employment Barriers - Pre-test (Time 1)
Description: Developed by Hong (2013). This is a 27-item self-report questionnaire that assesses the respondent's perception of employment barriers. It has the following subscales: Physical and mental health (6 items, scale range: 6-30), Labor Market Exclusion (3 items: scale range: 3 -15), Child Care (3 items: scale range: 3 -15). Human Capital (5 items, scale range: 5-25), and Soft Skills (5 items, scale range: 5-25). Higher scores represent higher/more barriers in that area.
Time Frame: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Childcare | 5.18 (3.37) | 4.86 (2.91)
  Human Capital | 9.86 (5.76) | 9.14 (4.89)
  Labor Market Exclusion | 5.47 (3.34) | 5.53 (3.26)
  Physical - Mental Health | 6.23 (4.53) | 5.71 (3.76)
  Soft Skill | 8.60 (5.38) | 8.50 (4.91)

47. Primary Outcome: Perceived Employment Barriers - Post--test (Time 2)
Description: as for outcome 46
Time Frame: Post-test (8weeks after pre-test/Time1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Childcare | 4.90 (3.26) | 5.04 (3.33)
  Human Capital | 9.03 (5.61) | 9.42 (5.68)
  Labor Market Exclusion | 4.68 (2.98) | 5.52 (3.35)
  Physical - Mental Health | 5.86 (4.21) | 5.86 (4.21)
  Soft Skill | 7.60 (4.80) | 8.39 (5.20)

48. Primary Outcome: Perceived Employment Barriers - Six-month Follow-up (Time 3)
Description: as for outcome 46
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Childcare | 4.18 (2.50) | 4.60 (2.96)
  Human Capital | 8.82 (5.07) | 8.36 (4.73)
  Labor Market Exclusion | 4.60 (2.75) | 5.25 (3.27)
  Physical - Mental Health | 5.74 (3.88) | 5.98 (4.33)
  Soft Skill | 8.25 (5.38) | 7.89 (4.78)

49. Primary Outcome: Employment Hope Scale - Pre-test (Time 1)
Description: Developed by Hong, Sheriff & Naeger, (2009) This is a 24-item self-report questionnaire that assesses the respondent's psychological readiness and hope for employment. Subscales included in the study are: Utilization Skills (4 items; scale range: 0-40); Self-Worth (4 items; scale range: 0-40); Self-Motivation (4 items; scale range: 0-40); Self-Perceived Capability (4 items; scale range: 0-40); Goal Orientation (4 items; scale range: 0-40); Future Job Outlook (4 items; scale range: 0-40); Psychological Empowerment (combined 12 items; scale range: 0-120); and Moving to Future Goals (combined 12 items; scale range: 0-120). Higher scores represent higher readiness or hope.
Time Frame: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Utilization Skills | 31.31 (10.80) | 32.01 (9.46)
  Self-Worth | 31.78 (10.01) | 31.67 (9.19)
  Psychological Empowerment | 92.40 (28.95) | 92.91 (26.39)
  Self-Motivation | 31.95 (10.42) | 32.60 (10.02)
  Self-Perceived Capability | 31.61 (10.09) | 31.54 (9.28)
  Moving to Future Goals | 92.60 (30.67) | 94.87 (27.04)
  Goal Orientation | 30.32 (10.86) | 31.26 (9.70)
  Future Job Outlook | 30.03 (10.33) | 31.00 (9.00)

50. Primary Outcome: Employment Hope Scale - Post-test (Time 2)
Description: as for outcome 49
Time Frame: Post-test (8weeks after pre-test/Time1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Utilization Skills | 32.01 (10.05) | 33.89 (8.50)
  Self-Worth | 31.91 (9.64) | 33.13 (8.58)
  Psychological Empowerment | 93.67 (28.15) | 97.42 (23.36)
  Self-Motivation | 32.60 (10.02) | 33.84 (8.53)
  Self-Perceived Capability | 31.88 (9.80) | 33.02 (8.14)
  Moving to Future Goals | 95.74 (28.99) | 98.25 (25.56)
  Goal Orientation | 31.84 (10.00) | 32.79 (8.68)
  Future Job Outlook | 30.81 (9.84) | 31.99 (8.81)

51. Primary Outcome: Employment Hope Scale - Six-month Follow-up (Time 3)
Description: as for outcome 49
Time Frame: Six-month follow up (six months after post-test/Time2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Utilization Skills | 29.84 (11.15) | 32.10 (8.75)
  Self-Worth | 29.27 (11.39) | 32.66 (8.60)
  Psychological Empowerment | 85.99 (32.31) | 94.19 (24.40)
  Self-Motivation | 29.33 (11.13) | 31.83 (9.07)
  Self-Perceived Capability | 29.06 (11.39) | 31.84 (8.39)
  Moving to Future Goals | 88.88 (32.04) | 94.93 (25.98)
  Goal Orientation | 29.83 (10.91) | 31.00 (8.92)
  Future Job Outlook | 28.34 (11.05) | 30.83 (8.71)

52. Other Pre Specified Outcome: Experiences in Close Relationships - Post-test (Time 2)
Description: Developed by Brennan, Clark, & Shaver (1998). This 36- item self report instrument measures avoidant and anxious attachment. Anxious scale has 18 items and avoidant scale has 18 items. Response answers range from 1 to 7. A total score for each subscale is calculated by adding the responses to each item and dividing it by the total number of. items. on the subscale So the total score for each subscale ranges from 1 to 7. Two total scores are calculated, one for each subscale. Higher scores represent more on that attachment dimension
Time Frame: Post-test (8 weeks after pre-test/Time1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 186 | 144
score on a scale
  Avoidance | 2.78 (1.08) | 2.52 (1.00)
  Anxiety | 3.14 (1.19) | 3.12 (1.23)

53. Other Pre Specified Outcome: Experience in Close Relationships - Pre-Test (Time 1)
Description: as for outcome 52
Time Frame: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 268 | 212
score on a scale
  Avoidance Subscale | 2.71 (1.05) | 2.67 (1.13)
  Anxiety Subscale | 3.20 (1.23) | 3.36 (1.16)

54. Other Pre Specified Outcome: Experiences in Close Relationships - Follow-up (Time 3)
Description: as for outcome 52
Time Frame: Follow-up (6 months after Post-test/Time2)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 118 | 96
score on a scale
  Avoidance | 2.76 (1.33) | 2.60 (0.90)
  Anxiety | 3.18 (1.26) | 3.01 (1.09)

ADVERSE EVENTS:
Time Frame: 8 to 10 months from Intake and Enrollment meeting until six-month follow-up (program exit). The range is due to the fact that for the intervention group couples could start their workshop one or two months after enrollment, then they would complete do the 8 week workshop (pre-test on first session and post- test on the last session) and then the six month follow-up (program exit).
Arm/Group | Control Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/290
Serious Adverse Events (participants affected / at risk) | 0/294 | 0/290
Other Adverse Events (participants affected / at risk) | 0/294 | 0/290

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT04227405/Prot_001.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT04227405/SAP_003.pdf
  • Informed Consent Form (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT04227405/ICF_002.pdf